CLINICAL TRIAL: NCT00016419
Title: A Phase II Study of Anti-Thymocyte Globulin and Cyclosporine for Patients With Myelodysplastic Syndrome (MDS)
Brief Title: S0020 Immunosuppressive Therapy in Treating Patients With Myelodysplastic Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S0020; S0020 (Other: SWOG); U10CA032102 (NIH)
Record Dates: First submitted 2001-05-06; First posted 2003-01-27 (Estimated); Last update posted 2015-03-06 (Estimated); Status verified 2015-03

CONDITIONS: Leukemia; Myelodysplastic Syndromes
Keywords: refractory anemia; refractory anemia with ringed sideroblasts; refractory anemia with excess blasts; de novo myelodysplastic syndromes; secondary myelodysplastic syndromes; childhood myelodysplastic syndromes
MeSH Terms: conditions — Leukemia; Myelodysplastic Syndromes; Anemia, Refractory; Anemia, Refractory, with Excess of Blasts | interventions — Antilymphocyte Serum; Cyclosporine

INTERVENTIONS:
Biological: anti-thymocyte globulin — 3.5 mg/kg/d IV over 12 hrs day 1
Drug: cyclosporine — 3 mg/kg bid days 5-94 then taper to 0 at day 124 PO

SUMMARY:
RATIONALE: Immunosuppressive therapy may improve bone marrow abnormalities and may be an effective treatment for myelodysplastic syndrome.

PURPOSE: Phase II trial to study the effectiveness of antithymocyte globulin plus cyclosporine in treating patients who have myelodysplastic syndrome.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the response in patients with myelodysplastic syndromes treated with anti-thymocyte globulin and cyclosporine.
* Determine the frequency and severity of toxic effects of this regimen in these patients.
* Assess the correlation between response to treatment and the in vitro assessment of T-lymphocyte subsets in these patients.

OUTLINE: This is a multicenter study. Patients are stratified according to myelodysplastic syndrome subclassification (refractory anemia [RA] vs RA with ringed sideroblasts vs RA with excess blasts).

Patients receive induction therapy comprising anti-thymocyte globulin IV over 6-12 hours on days 1-4 and oral cyclosporine twice daily on days 5-94 followed by a taper until day 124. Patients who relapse after a response of at least 60 days may receive reinduction therapy comprising oral cyclosporine twice daily on days 1-90 followed by a taper until day 120. Treatment continues in the absence of disease progression or unacceptable toxicity.

Patients are followed monthly for 6 months, every 2 months for 2 years, and then every 6 months for 3 years.

PROJECTED ACCRUAL: A total of 130 patients (53 with refractory anemia [RA], 33 with RA with ringed sideroblasts, and 44 with RA with excess blasts) will be accrued for this study within 14-22 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Morphologically confirmed myelodysplastic syndromes (MDS)

  * Refractory anemia (RA)
  * RA with ringed sideroblasts
  * RA with excess blasts
* Low, intermediate-1, or intermediate-2 risk by International Prognostic Scoring System criteria
* MDS secondary to prior chemotherapy and/or radiotherapy for other malignant disorders allowed
* Must have received prior transfusions of at least 4 units of red blood cells for anemia within the past 60 days
* Must be concurrently registered on SWOG-S9910 and SWOG-9007
* Ineligible for or refused participation in SWOG-S9920 (HLA-identical sibling peripheral blood stem cell transplantation)

PATIENT CHARACTERISTICS:

Age:

* 15 and over

Performance status:

* Zubrod 0-2

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Not specified

Other:

* No other malignancy within the past 2 years except adequately treated basal cell or squamous cell skin cancer, carcinoma in situ of the cervix, or adequately treated stage I or II cancer in complete remission
* HIV negative
* Not pregnant or nursing
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* See Disease Characteristics
* Prior cytokines (e.g., interferon or interleukin), colony-stimulating factors, or epoetin alfa allowed
* No prior bone marrow or stem cell transplantation
* No concurrent growth factors (including epoetin alfa) except filgrastim (G-CSF) or sargramostim (GM-CSF) for neutropenia

Chemotherapy:

* See Disease Characteristics
* No prior remission induction chemotherapy for MDS
* Prior hydroxyurea allowed

Endocrine therapy:

* Not specified

Radiotherapy:

* See Disease Characteristics

Surgery:

* Not specified

Other:

* Prior amifostine allowed
* No calcium-channel blockers (diltiazem, nicardipine, or verapamil), antifungals (fluconazole, itraconazole, or ketoconazole), antibiotics (clarithromycin or erythromycin), or other drugs (bromocriptine or danazol) that would increase cyclosporine concentrations for 48 hours before, during, and for 48 hours after cyclosporine
* No antibiotics (nafcillin or rifampin) or anticonvulsants (carbamazepine, phenobarbital, or phenytoin) that would decrease cyclosporine concentrations for 14 days before and during cyclosporine

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2001-08; Primary Completion 2003-07 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
total response | after induction therapy is completed

CONTACTS AND LOCATIONS:
Overall Officials: Charles A. Schiffer, MD, Study Chair — Barbara Ann Karmanos Cancer Institute
Locations (94):
- United States (94):
  - MBCCOP - Gulf Coast, Mobile, Alabama
  - CCOP - Greater Phoenix, Phoenix, Arizona
  - Veterans Affairs Medical Center - Phoenix (Carl T. Hayden), Phoenix, Arizona
  - Veterans Affairs Medical Center - Tucson, Tucson, Arizona
  - Arizona Cancer Center, Tucson, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Veterans Affairs Medical Center - Little Rock (McClellan), Little Rock, Arkansas
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - Veterans Affairs Medical Center - West Los Angeles, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Veterans Affairs Outpatient Clinic - Martinez, Martinez, California
  - CCOP - Bay Area Tumor Institute, Oakland, California
  - Chao Family Comprehensive Cancer Center, Orange, California
  - University of California Davis Cancer Center, Sacramento, California
  - CCOP - Santa Rosa Memorial Hospital, Santa Rosa, California
  - David Grant Medical Center, Travis Air Force Base, California
  - University of Colorado Cancer Center, Denver, Colorado
  - Veterans Affairs Medical Center - Denver, Denver, Colorado
  - MBCCOP - Howard University Cancer Center, Washington D.C., District of Columbia
  - CCOP - Atlanta Regional, Atlanta, Georgia
  - Dwight David Eisenhower Army Medical Center, Fort Gordon, Georgia
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - Tripler Army Medical Center, Honolulu, Hawaii
  - MBCCOP - University of Illinois at Chicago, Chicago, Illinois
  - Veterans Affairs Medical Center - Chicago (Westside Hospital), Chicago, Illinois
  - CCOP - Central Illinois, Decatur, Illinois
  - Veterans Affairs Medical Center - Hines (Hines Junior VA Hospital), Hines, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Genesis Medical Center, Davenport, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Veterans Affairs Medical Center - Wichita, Wichita, Kansas
  - Veterans Affairs Medical Center - Lexington, Lexington, Kentucky
  - Albert B. Chandler Medical Center, University of Kentucky, Lexington, Kentucky
  - MBCCOP - LSU Medical Center, New Orleans, Louisiana
  - Tulane University School of Medicine, New Orleans, Louisiana
  - Louisiana State University Health Sciences Center - Shreveport, Shreveport, Louisiana
  - Veterans Affairs Medical Center - Shreveport, Shreveport, Louisiana
  - Boston Medical Center, Boston, Massachusetts
  - Veterans Affairs Medical Center - Boston (Jamaica Plain), Jamaica Plain, Massachusetts
  - Veterans Affairs Medical Center - Ann Arbor, Ann Arbor, Michigan
  - CCOP - Ann Arbor Regional, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Veterans Affairs Medical Center - Detroit, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - CCOP - Grand Rapids, Grand Rapids, Michigan
  - CCOP - Beaumont, Royal Oak, Michigan
  - Providence Hospital - Southfield, Southfield, Michigan
  - Veterans Affairs Medical Center - Biloxi, Biloxi, Mississippi
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Veterans Affairs Medical Center - Jackson, Jackson, Mississippi
  - Keesler Medical Center - Keesler AFB, Keesler Air Force Base, Mississippi
  - Veterans Affairs Medical Center - Kansas City, Kansas City, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - St. Louis University Health Sciences Center, St Louis, Missouri
  - CCOP - St. Louis-Cape Girardeau, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Veterans Affairs Medical Center - Albuquerque, Albuquerque, New Mexico
  - MBCCOP - University of New Mexico HSC, Albuquerque, New Mexico
  - Veterans Affairs Medical Center - Albany, Albany, New York
  - Herbert Irving Comprehensive Cancer Center, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - CCOP - Southeast Cancer Control Consortium, Winston-Salem, North Carolina
  - Veterans Affairs Medical Center - Cincinnati, Cincinnati, Ohio
  - Barrett Cancer Center, Cincinnati, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Veterans Affairs Medical Center - Dayton, Dayton, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Veterans Affairs Medical Center - Oklahoma City, Oklahoma City, Oklahoma
  - Veterans Affairs Medical Center - Portland, Portland, Oregon
  - CCOP - Columbia River Program, Portland, Oregon
  - Oregon Cancer Institute, Portland, Oregon
  - Veterans Affairs Medical Center - Charleston, Charleston, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - CCOP - Greenville, Greenville, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - Veterans Affairs Medical Center - Houston, Houston, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Veterans Affairs Medical Center - San Antonio (Murphy), San Antonio, Texas
  - Veterans Affairs Medical Center - Temple, Temple, Texas
  - CCOP - Scott and White Hospital, Temple, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Veterans Affairs Medical Center - Salt Lake City, Salt Lake City, Utah
  - CCOP - Virginia Mason Research Center, Seattle, Washington
  - Veterans Affairs Medical Center - Seattle, Seattle, Washington
  - CCOP - Northwest, Tacoma, Washington
  - Madigan Army Medical Center, Tacoma, Washington